CLINICAL TRIAL: NCT04986358
Title: Short and Medium Term Postoperative Complications After Hallux Valgus Surgery
Acronym: HALLUXVALGUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Saint Jean, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LOCAL2021-WH01
Record Dates: First submitted 2021-07-22; First posted 2021-08-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-02

CONDITIONS: Hallux Valgus
Keywords: Hallux Valgus; Complications
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Intervention Model Description: Patient cohorte
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient cohorte (Other): Cohort of patients who will benefit from surgical management of their Hallux Valgus with post-operative follow-up at 2 years
  Interventions: Other: Follow up at 2 years

INTERVENTIONS:
Other: Follow up at 2 years — The patients will have a follow-up to carry out 2 years after their intervention in addition to their traditional care

SUMMARY:
The aim of this study is to make a precise inventory of the complications that may occur postoperatively in the more or less long term in a cohort of patients who should benefit from surgical management of Hallux Valgus.

DETAILED DESCRIPTION:
Hallux Valgus surgery is one of the most common foot surgeries. The surgical procedure itself has evolved a lot and is now, in almost all cases, on an outpatient basis with greatly improved pain management.

However, various postoperative complications, more or less severe and more or less long term, can worsen the final result. The literature describing these complications comes mainly from meta-analysis, retrospective studies or studies targeting a particular type of complications.

As a result, there are few complete and objective descriptions of these complications.

In addition, studies reporting postoperative consequences always assess the "serious" long-term complications responsible for a poor functional outcome, primarily the recurrence of the initial deformity, defined as surgical failure. It seemed relevant to try to assess early complications, "less serious", not necessarily worsening the final result but directly impacting the postoperative recovery period.

The evaluation of this recovery period and the length of time off work based on these "less severe" complications could improve the quality of surgical management of hallux valgus.

This is why it seemed interesting to carry out a precise inventory of the complications that may occur postoperatively in the more or less long term in a cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient with medical insurance.
* Patient who recieved information about study and signes a consent to participate in the study.
* Major patient requiring surgical management of a Hallux Valgus.

Exclusion Criteria:

* Minor patient.
* Patient participating in another interventional study.
* Patient with one of the following pathologies: Rheumatoid arthritis, haemophilia, inflammatory rheumatism or neurological spasticity.
* Patient to undergo a one-step bilateral Hallux Valgus surgical treatment (surgery of both feet on the same day).
* Patient refusing to sign the consent form.
* Patient for whom it is impossible to give informed information.
* Patient under the protection of justice, under curatorship ou under tutorship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2025-10-19 (Actual)

PRIMARY OUTCOMES:
Onset complication within 1 year after the intervention | 1 year
  Collection of the type of complication and its degree of severity (Clavien Dindo classification)

SECONDARY OUTCOMES:
Evaluation of patient satisfaction | 2 years
  satisfaction collected directly from the patient by a self-administered questionnaire : very satisfied, satisfied, not pronounced, dissatisfied or very dissatisfied.
Onset all complications within 2 years after the intervention | 2 years
  collection of the type of complication and its degree of severity (Clavien Dindo classification)

CONTACTS AND LOCATIONS:
Overall Officials: Wayan HEBRARD, MD, Principal Investigator — Clinique Saint Jean Sud de France
Locations (1):
- Clinique Saint Jean, Saint-Jean-de-Védas, France

REFERENCES:
- [Background] Monteagudo M, Martinez-de-Albornoz P. Management of Complications After Hallux Valgus Reconstruction. Foot Ankle Clin. 2020 Mar;25(1):151-167. doi: 10.1016/j.fcl.2019.10.011. Epub 2019 Nov 29. PMID 31997742
- [Background] Barg A, Harmer JR, Presson AP, Zhang C, Lackey M, Saltzman CL. Unfavorable Outcomes Following Surgical Treatment of Hallux Valgus Deformity: A Systematic Literature Review. J Bone Joint Surg Am. 2018 Sep 19;100(18):1563-1573. doi: 10.2106/JBJS.17.00975. PMID 30234626
- [Background] Raikin SM, Miller AG, Daniel J. Recurrence of hallux valgus: a review. Foot Ankle Clin. 2014 Jun;19(2):259-74. doi: 10.1016/j.fcl.2014.02.008. Epub 2014 Mar 29. PMID 24878414
- [Background] Filippi J, Briceno J. Complications after Metatarsal Osteotomies for Hallux Valgus: Malunion, Nonunion, Avascular Necrosis, and Metatarsophalangeal Osteoarthritis. Foot Ankle Clin. 2020 Mar;25(1):169-182. doi: 10.1016/j.fcl.2019.10.008. Epub 2019 Nov 26. PMID 31997743
- [Background] Lee KB, Kim MS, Park KS, Lee GW. Importance of postoperative sesamoid reduction on the outcomes of proximal chevron osteotomy for moderate to severe hallux valgus deformity. Foot Ankle Surg. 2019 Aug;25(4):434-440. doi: 10.1016/j.fas.2018.02.006. Epub 2018 Feb 16. PMID 30321971
- [Background] Lee KT, Park YU, Jegal H, Lee TH. Deceptions in hallux valgus: what to look for to limit failures. Foot Ankle Clin. 2014 Sep;19(3):361-70. doi: 10.1016/j.fcl.2014.06.003. Epub 2014 Jul 2. PMID 25129349
- [Background] Nix S, Smith M, Vicenzino B. Prevalence of hallux valgus in the general population: a systematic review and meta-analysis. J Foot Ankle Res. 2010 Sep 27;3:21. doi: 10.1186/1757-1146-3-21. PMID 20868524
- [Background] Zambelli R, Baumfeld D. Intraoperative and Postoperative Evaluation of Hallux Valgus Correction: What Is Important? Foot Ankle Clin. 2020 Mar;25(1):127-139. doi: 10.1016/j.fcl.2019.10.007. Epub 2019 Dec 4. PMID 31997740
- [Background] Bock P, Kluger R, Kristen KH, Mittlbock M, Schuh R, Trnka HJ. The Scarf Osteotomy with Minimally Invasive Lateral Release for Treatment of Hallux Valgus Deformity: Intermediate and Long-Term Results. J Bone Joint Surg Am. 2015 Aug 5;97(15):1238-45. doi: 10.2106/JBJS.N.00971. PMID 26246258
- [Background] Jeuken RM, Schotanus MG, Kort NP, Deenik A, Jong B, Hendrickx RP. Long-term Follow-up of a Randomized Controlled Trial Comparing Scarf to Chevron Osteotomy in Hallux Valgus Correction. Foot Ankle Int. 2016 Jul;37(7):687-95. doi: 10.1177/1071100716639574. Epub 2016 Mar 23. PMID 27009063
- [Background] Lee KB, Cho NY, Park HW, Seon JK, Lee SH. A comparison of proximal and distal Chevron osteotomy, both with lateral soft-tissue release, for moderate to severe hallux valgus in patients undergoing simultaneous bilateral correction: a prospective randomised controlled trial. Bone Joint J. 2015 Feb;97-B(2):202-7. doi: 10.1302/0301-620X.97B2.34449. PMID 25628283
- [Background] Lai MC, Rikhraj IS, Woo YL, Yeo W, Ng YCS, Koo K. Clinical and Radiological Outcomes Comparing Percutaneous Chevron-Akin Osteotomies vs Open Scarf-Akin Osteotomies for Hallux Valgus. Foot Ankle Int. 2018 Mar;39(3):311-317. doi: 10.1177/1071100717745282. Epub 2017 Dec 14. PMID 29241361
- [Background] Brogan K, Lindisfarne E, Akehurst H, Farook U, Shrier W, Palmer S. Minimally Invasive and Open Distal Chevron Osteotomy for Mild to Moderate Hallux Valgus. Foot Ankle Int. 2016 Nov;37(11):1197-1204. doi: 10.1177/1071100716656440. Epub 2016 Jul 4. PMID 27381179
- [Background] Kaufmann G, Mortlbauer L, Hofer-Picout P, Dammerer D, Ban M, Liebensteiner M. Five-Year Follow-up of Minimally Invasive Distal Metatarsal Chevron Osteotomy in Comparison with the Open Technique: A Randomized Controlled Trial. J Bone Joint Surg Am. 2020 May 20;102(10):873-879. doi: 10.2106/JBJS.19.00981. PMID 32149929
- [Background] Chong A, Nazarian N, Chandrananth J, Tacey M, Shepherd D, Tran P. Surgery for the correction of hallux valgus: minimum five-year results with a validated patient-reported outcome tool and regression analysis. Bone Joint J. 2015 Feb;97-B(2):208-14. doi: 10.1302/0301-620X.97B2.34891. PMID 25628284
- [Background] Dawson J, Boller I, Doll H, Lavis G, Sharp R, Cooke P, Jenkinson C. Responsiveness of the Manchester-Oxford Foot Questionnaire (MOXFQ) compared with AOFAS, SF-36 and EQ-5D assessments following foot or ankle surgery. J Bone Joint Surg Br. 2012 Feb;94(2):215-21. doi: 10.1302/0301-620X.94B2.27634. PMID 22323689
- [Background] Coughlin MJ, Freund E. Roger A. Mann Award . The reliability of angular measurements in hallux valgus deformities. Foot Ankle Int. 2001 May;22(5):369-79. doi: 10.1177/107110070102200503. PMID 11428754
- [Background] Lee KM, Ahn S, Chung CY, Sung KH, Park MS. Reliability and relationship of radiographic measurements in hallux valgus. Clin Orthop Relat Res. 2012 Sep;470(9):2613-21. doi: 10.1007/s11999-012-2368-6. Epub 2012 Apr 28. PMID 22544667
- [Background] Talbot KD, Saltzman CL. Assessing sesamoid subluxation: how good is the AP radiograph? Foot Ankle Int. 1998 Aug;19(8):547-54. doi: 10.1177/107110079801900808. PMID 9728703
- [Background] Smith RW, Reynolds JC, Stewart MJ. Hallux valgus assessment: report of research committee of American Orthopaedic Foot and Ankle Society. Foot Ankle. 1984 Sep-Oct;5(2):92-103. doi: 10.1177/107110078400500208. No abstract available. PMID 6389278
- [Background] Coughlin MJ. Hallux valgus. J Bone Joint Surg Am. 1996 Jun;78(6):932-66. No abstract available. PMID 8666613
- [Background] Lewis TL, Ray R, Miller G, Gordon DJ. Third-Generation Minimally Invasive Chevron and Akin Osteotomies (MICA) in Hallux Valgus Surgery: Two-Year Follow-up of 292 Cases. J Bone Joint Surg Am. 2021 Jul 7;103(13):1203-1211. doi: 10.2106/JBJS.20.01178. PMID 33764936
- [Background] Lehman DE. Salvage of complications of hallux valgus surgery. Foot Ankle Clin. 2003 Mar;8(1):15-35. doi: 10.1016/s1083-7515(02)00130-4. PMID 12760572
- [Background] Costa MT, de Almeida Pinto RZ, Ferreira RC, Sakata MA, Frizzo GG, Santin RA. OSTEOTOMY OF THE FIRST METATARSAL BASE ON THE TREATMENT OF MODERATE TO SEVERE HALLUX VALGUS RESULTS AFTER MEAN FOLLOW-UP TIME OF EIGHT YEARS. Rev Bras Ortop. 2015 Nov 16;44(3):247-53. doi: 10.1016/S2255-4971(15)30075-6. eCollection 2009 Jan. PMID 27004179
- [Background] Fuhrmann RA, Zollinger-Kies H, Kundert HP. Mid-term results of Scarf osteotomy in hallux valgus. Int Orthop. 2010 Oct;34(7):981-9. doi: 10.1007/s00264-010-0958-z. Epub 2010 Feb 16. PMID 20157812